CLINICAL TRIAL: NCT06064344
Title: Safety and Efficacy of Intralesional Rituximab Injection Versus Involved Site Radiation Therapy in Primary Ocular Adnexal MALT Lymphoma: a Multicenter Non-Inferiority Randomized Controlled Trial
Brief Title: RCT of Intralesional Rituximab Injection Versus Involved Site Radiation Therapy in Ocular Adnexal MALT Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong Lu, Professor, MD, PhD, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023KYPJ125
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Primary Ocular Adnexal MALT Lymphoma
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional Rituximab Injection (Experimental)
  Interventions: Drug: Rituximab
- Involved Site Radiation Therapy (Active Comparator)
  Interventions: Radiation: Involved Site Radiation Therapy

INTERVENTIONS:
Drug: Rituximab — Intralesional Rituximab Injection
  Arms: Intralesional Rituximab Injection
Radiation: Involved Site Radiation Therapy — Involved Site Radiation Therapy
  Arms: Involved Site Radiation Therapy

SUMMARY:
This project proposes to establish a prospective, multicenter, randomized, controlled clinical study to compare the safety and efficacy of Intralesional Rituximab Injection versus Involved Site Radiation Therapy for the treatment of primary ocular adnexal MALT lymphoma. The aim is to provide high-level clinical evidence for the treatment of ocular adnexal MALT lymphoma and to offer patients treatment options that have fewer complications and comparable therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old.
2. Meets the WHO diagnostic criteria for ocular adnexal MALT lymphoma, with a comprehensive diagnosis based on pathology (including pathological morphology, immunophenotype, and genetic testing), clinical manifestations, and biological characteristics:

   1. Clinical criteria: ① Extranodal lymphoma occurring in the ocular adnexa; ② Localized mass.
   2. Pathological criteria:

   <!-- -->

   1. Histopathology: Morphological features that recapitulate Peyer's patches, including: ① Lymphoepithelial lesions; ② Reactive follicles; ③ Marginal zone cells and/or monocytoid B cells; ④ Small lymphocyte-like cells; ⑤ Plasma cells; ⑥ Scattered transformed blasts (centroblast-like, immunoblast-like cells).
   2. Immunophenotype: Tumor cells express B-cell-related antigens: SIgM+, CIg +/-, CD5-, CD10-, CD23-, cyclin DI, CD43 +/-, CD19, CD20, CD22, and CD79a positive.
   3. Genetic features: Absence of BCL-1 and BCL-2 gene rearrangements, presence of IgH/L gene rearrangements; possible +3 and t(11, 18)(q21, q21).
3. Based on the TNM staging of ocular adnexal lymphoma, patients with stages T1-3 of ocular adnexal MALT lymphoma are included.
4. Informed and signed informed consent.

Exclusion Criteria:

1. Based on the TNM staging of ocular adnexal lymphoma, patients staged as T4 of ocular adnexal MALT lymphoma.
2. Patients who have previously received local or systemic radiation, chemotherapy, or drug treatment specifically for ocular adnexal MALT lymphoma.
3. Presence of cataract and is anticipated to require surgical treatment within a certain period after enrollment; existing cataract affects visual field testing and fundoscopic examination; vision affected by cataract is <20/40.
4. In addition to the need for treatment of ocular adnexal MALT lymphoma, there is a requirement for other ocular procedures (e.g., full-thickness corneal transplant or retinal surgery) or an anticipated need for another emergent ocular surgery.
5. Concurrent other ocular diseases: Including corneal abnormalities or existing corneal infections, iridocorneal endothelial syndrome, anterior segment dysgenesis, true microphthalmos, uveitis, glaucoma, ocular trauma, and retinal disorders such as central retinal vein occlusion, central retinal artery occlusion, retinal detachment, etc.
6. Need for long-term use of local or systemic steroids.
7. Patients already enrolled in other drug clinical trials.
8. Pregnant or breastfeeding women.
9. Serious systemic diseases: Advanced cardiac disease, kidney disease, respiratory diseases, or other malignant tumors, etc.
10. Inability to understand the research content.

If both eyes of a patient meet the inclusion criteria, the right eye will be selected for participation in the study, while the left eye will receive the same treatment, but its data will not be included in the research. Each patient can have only one eye participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-10-07 (Estimated); Primary Completion 2027-10-06 (Estimated); Study Completion 2027-10-06 (Estimated)

PRIMARY OUTCOMES:
The cumulative occurrence rate of complications of grade ≥2 within 2 years after the start of treatment | 2 years after the start of treatment

SECONDARY OUTCOMES:
Local control rate of ocular adnexal MALT lymphoma 2 years after the start of treatment | 2 years after the start of treatment
2-year Time-to-next-treatment rate | 2 years after the start of treatment
2-year overall survival rate | 2 years after the start of treatment

IPD SHARING:
Plan to Share IPD: No